CLINICAL TRIAL: NCT05949203
Title: Oregon PrEP at Home Study: Real-world Delivery of Long-acting Cabotegravir (CAB-LA) for HIV Pre-exposure Prophylaxis (PrEP) Through a Tele-PrEP Program and a Home Infusion Program Partnership to Address Geographic PrEP Disparities in Oregon
Brief Title: Oregon PrEP at Home Study
Acronym: OR-PrEP@Home
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: STUDY00025207
Record Dates: First submitted 2023-06-26; First posted 2023-07-17 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-06

CONDITIONS: HIV/AIDS
Keywords: HIV prevention; PrEP; telemedicine; home infusion pharmacy; long-acting cabotegravir
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — cabotegravir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All participants: All participants will receive standard-of-care through the tele-PrEP program and home infusion pharmacy.
  Interventions: Drug: Cabotegravir Injection

INTERVENTIONS:
Drug: Cabotegravir Injection — Administration of HIV pre-exposure prophylaxis with cabotegravir 600 mg/3mL extended release injectable suspension every other month.
  Other Names: Apretude

SUMMARY:
This demonstration study will evaluate the real-world implementation of long-acting cabotegravir (CAB-LA) for HIV pre-exposure prevention (PrEP) through a partnership between the OHSU Tele-PrEP Program (TPP) and the OHSU Home Infusion Pharmacy (HIP). The study will perform a formative evaluation of the TPP/HIP partnership to determine its merit and worth, with revisions made as needed to improve the program, which is reflective of a real-world program rollout. The study is observational, and there is no comparison group. The primary objective is to evaluate adherence to CAB-LA by both urban and rural participants using the TPP/HIP partnership. The goals of the study are improve the TPP/HIP program itself with attention to reducing geographic disparities, and to disseminate best practices and lessons learned to the broader HIV prevention community.

ELIGIBILITY:
Inclusion Criteria:

* Residence in Oregon
* English or Spanish spoken and written language ability
* Clinical eligibility for PrEP with CAB-LA including HIV-negative serostatus
* Access to stable Internet
* Access to a clean, safe location that is appropriate for home administration

Exclusion Criteria:

* Clinical ineligibility for PrEP with CAB-LA including HIV-positive serostatus, injection drug use as only HIV risk factor, or clinical contraindication (such as a hypersensitivity reaction to CAB-LA or use of a contraindicated medication).
* Uninsured
* Payer does not cover HIP services
* Pregnancy
* Residence outside of the home infusion program's catchment area
* Incarceration
* Decisional impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All genders are eligible
Study Population: Residents of Oregon age 18 or older who are eligible for HIV pre-exposure prophylaxis with long-acting cabotegravir through the OHSU Tele-PrEP Program and OHSU Home Infusion Pharmacy. People of childbearing potential or who are breast/chest feeding are eligible, but pregnant people are ineligible.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
On-time initiation and continuation doses | 24 months
  Proportion of on-time initiation and continuation doses of CAB-LA administered

SECONDARY OUTCOMES:
Successful home infusion pharmacy referrals | 24 months
  Proportion of referrals to home infusion that result in successful CAB-LA initiation over the study period
Time to initiation | 24 months
  Time in days between first tele-PrEP appointment and administration of first CAB-LA dose
Persistence rate | 24 months
  The persistence rate of participation in the tele-PrEP/home infusion pharmacy program for administration of CAB-LA
Sexually transmitted infection screenings | 24 months
  Number of HIV, gonorrhea, chlamydia, and syphilis screenings per participant over 10 months of CAB-LA continuation
Participant experience | 24 months
  Assessment of TPP/HIP program for delivery of CAB-LA continuation therapy using a bespoke questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher B Fox, MSN, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data and adverse event reporting will be shared with the study partner ViiV Healthcare.